CLINICAL TRIAL: NCT02945748
Title: Uninvasive Cardiac Output Monitoring (USCOM) in Critically Ill Children: Validation and Prediction of Hemodynamic Instability
Status: Completed | Type: Observational
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 0693-14-RMC
Record Dates: First submitted 2016-10-25; First posted 2016-10-26 (Estimated); Last update posted 2021-03-16 (Actual); Status verified 2020-08

CONDITIONS: Hemodynamic Instability
Keywords: pediatric; cardiac output; fluid responsiveness; critically ill; hemodynamic monitoring
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Hemodynamically unstable ventilated PICU & PCICU patients, which a decision for commencement in inotropic therapy or fluid bolus has been made, will be recruited. Hemodynamic measurements will be carried out before and after therapy have been made, including customary hemodynamic parameters, echocardiography and USCOM studies.

All parameters will be analyzed for fluid responsiveness or inotropic therapy prediction. Trend in USCOM parameters will be compared to echocardiography CO parameters.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric critically ill ventilated patients admitted to PICU & PCICU
* Hemodynamically unstable which a decision for commencement in inotropic therapy or fluid bolus has been made
* parental concent

Exclusion Criteria:

* Cardiac shunt
* Aortal anomaly \ Repair
* Tracheostomy
* Parental refusal to participate

Ages: 2 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric critically ill ventilated patients addmited to PICU & PCICU
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2016-07; Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Raise>10% in cardiac index following therapy | 20 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Schneider's children medical center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No